CLINICAL TRIAL: NCT02597192
Title: Professor Doctor, Cukurova University Faculty of Dentistry
Brief Title: Clinical Effects of Bacillus Containing Oral Hygiene Products on Gingivitis: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Onur Ozcelik, Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CukurovaU-7
Record Dates: First submitted 2015-10-30; First posted 2015-11-05 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Gingivitis
Keywords: gingivitis; gingival inflammation; probiotics; Bacillus
MeSH Terms: conditions — Gingivitis | interventions — PIP protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active test group (Active Comparator): probiotic oral hygiene products with Bacillus (PIP, Chrisal)
  Interventions: Other: probiotic oral hygiene products with Bacillus (PIP, Chrisal)
- Placebo group (Placebo Comparator): oral hygiene products without Bacillus
  Interventions: Other: oral hygiene products without Bacillus

INTERVENTIONS:
Other: probiotic oral hygiene products with Bacillus (PIP, Chrisal) — products with Bacillus probiotics
  Arms: Active test group
Other: oral hygiene products without Bacillus — products without Bacillus
  Arms: Placebo group

SUMMARY:
Aim: Evaluating the clinical effects of a Bacillus subtilis, Bacillus megaterium and Bacillus pumulus containing toothpaste, mouthwash and toothbrush cleaner versus a placebo in patients with generalized gingivitis.

Materials and methods: In this double-blind placebo-controlled randomized clinical trial generalized gingivitis patients who were systemically healthy and who did not smoke were included. They used a placebo or probiotic Bacillus containing toothbrush cleaner for 8 weeks. Primary outcome measures of interest were plaque and gingivitis index, secondary outcome measures were pocket probing depth and bleeding on probing.

DETAILED DESCRIPTION:
The administration of micro-organisms to improve the human health was already promoted by the Nobel prizewinning scientist Eli Metchnikoff in the beginning of the 20th century. However, it took several decades for this subject to become a topic of interest in medicine. At this moment these micro-organisms are called "probiotics" and defined as "living microorganisms which, when administered in adequate amounts, confer a health benefit for the host" (http://www.who.int/foodsafety/publications/fs_management/en/probiotics.pdf). Over the past decade probiotics have been extensively investigated from the perspective of oral health. It was shown that probiotics have the capacity to reduce mutans streptococci counts in saliva and/or plaque during their usage, that they have a positive influence on bad breath and that they can improve the results of scaling and root planing in periodontitis patients. A positive effect of probiotic usage on plaque accumulation and gingivitis measurements in gingivitis patients was also shown.To the investigators knowledge, at this moment no trials are available describing the effect of other probiotic genera on gingivitis. Since it is clear that probiotic effects are strain, dosage and mode of application dependent, the aim of this study was to evaluate the use of a probiotic toothpaste, mouthwash and toothbrush cleaner with Bacillus subtilis, Bacillus megaterium, and Bacillus pumulus versus a placebo in patients with generalized gingivitis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with plaque-induced gingivitis
* a pocket probing depth not more than 5 mm
* at least 20 natural teeth
* no history of periodontal therapy or previous use of antibiotics or anti-inflammatory medication within the preceding 6 months

Exclusion Criteria:

* patients with hematologic disorders, or other systemic illness
* pregnant and lactating females
* patients undergoing orthodontic treatment
* those with smoking habits were excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
gingival index scores | 8weeks

SECONDARY OUTCOMES:
plaque index scores | 8weeks

CONTACTS AND LOCATIONS:
Overall Officials: Onur Ozcelik, Professor, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)